CLINICAL TRIAL: NCT02723097
Title: A Pilot Test of the Relaxation Response Resiliency Program (3RP) in Spanish Speaking World Trade Center Survivors With Post Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-00721
Record Dates: First submitted 2016-03-24; First posted 2016-03-30 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Post Traumatic Stress Disorder (PTSD)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Relaxation Response Resiliency Program (3RP) (Experimental)
  Interventions: Behavioral: 3 RP

INTERVENTIONS:
Behavioral: 3 RP
  Other Names: Relaxation Response Resiliency Program

SUMMARY:
The objective of this protocol is to test the feasibility and acceptability of the Relaxation Response Resiliency Program (3RP), a psychotherapy treatment providing a variety of mind body skills and interventions to decrease medical and mental health symptoms and build resilience, in Spanish-speaking World Trade Center (WTC) survivors, and to examine its clinical effectiveness to reduce Post Traumatic Stress Disorder (PTSD), depression, anxiety, and lower respiratory symptoms (LRS) and improve psychosocial functioning.

ELIGIBILITY:
Inclusion Criteria:

* score > or = 44 on the PTSD Checklist PCL, considered the broad definition of PTSD syndrome71
* report at least one LRS symptoms (i.e., shortness of breath, wheezing, dyspnea or cough).
* Spanish Speaking

Exclusion Criteria:

* regular practice of eliciting relaxation response (i.e., meditation, yoga) in the past 6 months,
* serious unmanaged mental illness including bipolar disorder, psychosis, and active substance misuse disorders;
* inability to participate in consecutive sessions over 3-month period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-10-11 (Actual); Study Completion 2017-10-11 (Actual)

PRIMARY OUTCOMES:
Structured Clinical Interview (SCID-NP) for Diagnostic and Statistical Manual DSM-IV | 1 Month
  State-of-the-art instrument for obtaining psychiatric diagnoses.
Symptom Severity using PTSD Checklist | 1 Month
  Symptoms will be assessed with the PTSD Checklist (PCL), a 17-item self-report measure of current (past month) PTSD symptoms based on the DSM-IV criteria. It is a widely-used and validated measure of PTSD symptom severity.
Assessment of Anxiety Symptoms using Generalized Anxiety Disorder Scale (GAD-7) | 1 Month
Measure of Functional Impairment using the Range of Impaired Functioning Tool (RIFT) | 1 Month
  widely-used instrument that taps the domains of work, household duties, interpersonal relationships, recreation, and subjective satisfaction with life. Each domain is rated on a five-point scale from very good to very poor. The total score is the sum of the different domains.
Assessment of Mindful attention using Mindful Attention Awareness Scale (MAAS) | 1 Month
  The MAAS is a 15-item questionnaire on which respondents indicate, on a 6 point Likert-type scale (1 = almost always to 6 = almost never), their level of awareness and attention to present events and experiences.
Health Promoting Behaviors will be assessed with the Health Promoting Lifestyles Profile-II (HPLP-II) | 1 Month
  he HPLP-II is a 52 item self-report inventory of health behaviors and has been used in previous mind-body treatment studies
Measure of treatment expectancy using the Treatment Credibility/Expectancy Questionnaire. | 1 Month
  The 6-item Treatment Credibility/Expectancy Questionnaire (CEQ)84 will be used to examine treatment expectancy related to the 3RP.

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Ferri, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States